CLINICAL TRIAL: NCT03711214
Title: Analysis of the Immune Profile of Saliva and Serum of Patients With Primary Sjögren´s Syndrome
Brief Title: Immune Profile of Saliva and Serum of Patients With Primary Sjögren´s Syndrome
Acronym: pSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPS - pSS; 2015/03756-4 (Other Grant/Funding Number: FAPESP); 2018/09937-9 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2018-09-03; First posted 2018-10-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Clinical treatment of periodontal disease in pSS patients and healthy individuals
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pSS patients (Active Comparator): We will evaluate 40 patients with pSS (EULAR/ACR Classification Criteria, 2016) of both sexes before and after periodontal disease treatment.
  Interventions: Procedure: Periodontal scaling
- Healthy individuals (Active Comparator): We will evaluate 40 healthy controls before and after periodontal disease treatment.
  Interventions: Procedure: Periodontal scaling

INTERVENTIONS:
Procedure: Periodontal scaling — Periodontal scaling and root planing
  Other Names: Clinical periodontal disease treatment

SUMMARY:
Primary Sjögren's syndrome (pSS) is a chronic systemic inflammatory disease, which mainly affects the lacrimal and salivary glands, leading to sicca syndrome. pSS has a probable autoimmune etiology, with the production of several autoantibodies such as antinuclear antibodies (ANA), anti-Ro/SS-A, anti-La/SS-B, rheumatoid factor (RF) and cryoglobulins. Recently, our group described a high frequency of antibodies directed to DNase I in the serum of pSS patients and these antibodies were associated with the presence of the anti-Epstein-Barr (EBV) early antigen diffuse (anti-EA-D). This finding becomes interesting considering the recent description of reduction of DNase I activity in the tear of patients with xerophthalmia of different causes, which would result in an accumulation of extracellular DNA and neutrophilic inflammatory infiltrate on the ocular surface. This hypothesis is reinforced by the observation that treatment with DNase I as eye drops results in clinical improvement of dry eye. In addition, it has been shown that periodontal disease is an aggravating factor of xerostomia in pSS, as it leads to a chronic inflammatory process and, consequently, to the destruction of minor salivary glands. Therefore, the objective of the present study will be to evaluate the presence of antibodies directed to DNase I in the saliva and serum of pSS patients and its possible capacity of inhibition of the enzyme before and after treatment of periodontal disease. Such findings will be correlated with the presence of periodontal disease, with the glandular and extraglandular manifestations of SSp and also with the presence of EBV DNA in the serum and oral lavage of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary Sjögren's syndrome according to 2016 EULAR/ACR Classification Criteria, and healthy people without any rheumatic disease/symptoms of sicca syndrome
* Patients regularly followed at the Sjögren's Syndrome outpatient clinic of Rheumatology Division

Exclusion Criteria:

* Use of drugs that cause oral dryness (mainly antidepressants and antihistamines).
* Patients with history of head and neck radiation therapy.
* Current smoking.
* Pregnancy and/or lactation.
* History of periodontal treatment for at least 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Xerostomia Inventory Score at 3 months | Change from baseline Xerostomia Inventory Score at 3 months
  Change from baseline Xerostomia Inventory Score at 3 months. An international validated questionnaire of dry mouth symptoms ranging from 11 to 55 points.
Change from baseline activity of DNAse I enzyme in saliva at 3 months | Change from baseline activity of DNAse I enzyme in saliva at 3 months
  Change from baseline activity of DNAse I enzyme in saliva at 3 months measured by Enzyme-Linked Immunosorbent Assay (ELISA).

SECONDARY OUTCOMES:
Change from baseline interleukin-1b (IL-1b) concentration in saliva at 3 months | Change from baseline interleukin-1b (IL-1b) concentration in saliva at 3 months
  Change from baseline interleukin-1b (IL-1b) concentration in saliva at 3 months measured by Luminex Assay.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrosio LM, Rovai ES, Franca BN, Balzarini DA, Abreu IS, Lopes SB, Nunes TB, Lourenco SV, Pasoto SG, Saraiva L, Holzhausen M. Effects of periodontal treatment on primary sjogren's syndrome symptoms. Braz Oral Res. 2017 Jan 16;31:e8. doi: 10.1590/1807-3107BOR-2017.vol31.0008. PMID 28099577
- [Background] Nakamura-Kiyama M, Ono K, Masuda W, Hitomi S, Matsuo K, Usui M, Nakashima K, Yokota M, Inenaga K. Changes of salivary functions in experimental periodontitis model rats. Arch Oral Biol. 2014 Feb;59(2):125-32. doi: 10.1016/j.archoralbio.2013.11.001. Epub 2013 Nov 8. PMID 24370183
- [Derived] Martins VAO, Floriano TF, Leon EP, Villamarin LEB, Deveza GBH, Aikawa NE, Silva CAA, Kupa LVK, Peres MPSM, Braz-Silva PH, Bonfa E, Pasoto SG. Primary dental care treatment in primary Sjogren's syndrome: a possible role in improving salivary flow rate. Clin Exp Rheumatol. 2022 Dec;40(12):2258-2267. doi: 10.55563/clinexprheumatol/kfn28h. Epub 2022 Sep 26. PMID 36189908